CLINICAL TRIAL: NCT00000156
Title: The Effects of Light Reduction on Retinopathy of Prematurity (Light-ROP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-58
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2006-06-05 (Estimated); Status verified 2003-10

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Eye Protective Devices

INTERVENTIONS:
Device: Goggles
Procedure: Ambient Light Reduction

SUMMARY:
To evaluate the effect of ambient light reduction on the incidence of retinopathy of prematurity (ROP).

DETAILED DESCRIPTION:
Despite progress during the past decade in treatment of ROP, this disease still poses a significant (approximately 2.1 percent) risk of blindness to extremely low birth-weight (<1,251 grams) preterm infants. Current estimates indicate that about 27,000 infants of extremely low birth weight are born annually, of which 74 percent will survive. As techniques of managing smaller and less mature preterm infants continue to improve, it is expected that the number of infants at risk for blindness will continue to increase.

For infants weighing less than 1,251 grams at birth, the Cryotherapy for Retinopathy of Prematurity (CRYO-ROP) Study has shown that the risk of developing severe, acute (threshold) ROP is 6 percent. Although cryotherapy, when applied at the time of threshold ROP, reduces the rate of unfavorable visual outcome, 35 percent of eyes that develop this level of severe, acute disease are blind 1 year after treatment. Moreover, cryotherapy is destructive. Even when cryotherapy prevents progression to retinal detachment, it is associated with peripheral retinal destruction and may, in some cases, be associated with subnormal central vision due to high myopia and/or macular scarring. Corrective surgical treatments for retinal detachment caused by ROP have proven to be of little visual benefit. A preventive treatment for ROP that is safe, efficacious, easily applied, and inexpensive is desirable.

The investigators hypothesize that reducing the amount of light that reaches the eyes of preterm infants may be effective in preventing ROP. Although previous reports on the use of light reduction to the eyes of preterm infants in the nursery have produced conflicting results, there are sufficient reasons to believe that this strategy may be effective in reducing the incidence and severity of ROP. These reasons center on the role of light in the production of destructive free radicals. Supplemental oxygen produces the same free radicals, and the two mechanisms may be additive.

In this masked, controlled study, infants weighing less than 1,251 grams at birth were prospectively randomized within 24 hours of birth to wear goggles or not to wear goggles. Goggles contain 97 percent near neutral density filters and were worn until the infant reached either 31 weeks gestational age or 4 weeks postnatal age, whichever was longer. The goggled and nongoggled infants were exposed to the same ambient light conditions within any given Study Center. Eyes of all infants were examined on a prescribed schedule by certified examiners to determine the incidence of any confirmed ROP.

The primary objective of this study is to answer the following question: Does light reduction to the eyes of extremely low birth-weight infants decrease the incidence of any confirmed ROP (at least 3 contiguous clock hours, any stage, any zone)? The primary end points are therefore ROP or full vascularization.

The secondary objective of this study is to evaluate the following question: Does light reduction to the eyes of extremely low birth-weight infants decrease the incidence of more severe ROP (prethreshold ROP -- the secondary end point)?

The study has recruited approximately 400 infants, equally divided into goggle-wearing and control group. Since randomization must occur within 24 hours of birth, the investigators anticipate a mortality rate of between 10 percent and 20 percent of enrollees prior to outcome. The study is in the followup phase with regular ophthalmologic exams until either ROP regression or normal full retinal vascularization is established. A final exam occurs at adjusted age 6 months.

ELIGIBILITY:
Premature infants weighing less than 1,251 grams at birth and having a gestational age of less than 31 weeks were eligible for randomization. Consent must have been obtained within 24 hours of birth. Patients with major congenital anomalies are excluded.

Max Age: 1 Day | Sex: All
Age Groups: Child
Dates: Start 1995-07

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Children's Hospital of Buffalo, Buffalo, New York
  - The University of Texas, Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas, Health Science Center, San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Reynolds JD, Hardy RJ, Kennedy KA, Spencer R, van Heuven WA, Fielder AR. Lack of efficacy of light reduction in preventing retinopathy of prematurity. Light Reduction in Retinopathy of Prematurity (LIGHT-ROP) Cooperative Group. N Engl J Med. 1998 May 28;338(22):1572-6. doi: 10.1056/NEJM199805283382202. PMID 9603794